CLINICAL TRIAL: NCT00518570
Title: A Pilot Study: Levetiracetam in the Treatment of Patients With Premenstrual Dysphoric Disorder
Brief Title: Levetiracetam in the Treatment of Patients With Premenstrual Dysphoric Disorder (PMDD)
Acronym: pmdd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berkshire Health Systems (Other)
Collaborators: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Levetiracetam and PMDD; BMC03-010
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2007-08-20 (Estimated); Status verified 2007-08

CONDITIONS: Premenstrual Dysphoric Disorder
Keywords: PMDD; PMS; Levetiracetam
MeSH Terms: conditions — Premenstrual Dysphoric Disorder | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label treatment (Experimental): Patients prospectively diagnosed with premenstrual dysphoric disorder.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam was started at 250 mg qhs at the end of the first week of the follicular phase. Dose was gradually increased up to 1500 mg bid as tolerated or clinically effective. The treatment phase lasted 4 months.
  Other Names: Keppra

SUMMARY:
The purpose of this study is to investigate the clinical efficacy of Levetiracetam in the treatment of symptoms of premenstrual dysphoric disorder (PMDD) in an open label study.

ELIGIBILITY:
Inclusion Criteria:

PMDD diagnostic and severity criteria:

1. Women with PMDD according to DSM-IV-TR criteria

   * At screening by history
   * At the end of the Qualification Phase by review of symptom records.
2. The first 2 consecutive or 2 out of 3 consecutive qualification cycles must fulfill the following criteria:

   * For women who were not on any medications for the PMDD symptoms:

     * Late luteal phase (7 days which include the last six days before menses through day one) daily average of > or equal 3.5 for at least 4 of 7 of these days on any 5 distinct items with no overlap on Daily Record of Severity of Problems (DRSP) Scale, at least one item must represent a non-physical symptom. Entries in the diary must be present for at least three of these days for the item to be used as an inclusion criterion for that month.
     * Follicular phase (days 8-12 after first day of menses) daily average less than or equal 2.5 on DRSP scale for non-physical symptoms only. The average will be calculated for days 8-12 of the cycle, day 1 being the first day of menstrual bleeding. Entries in the diary must be present for at least three of these days for the item to be used as an inclusion criterion for that month.
     * Late luteal phase (6 days before menses through day 1) daily average at least twice as high as follicular phase daily average for five distinct items.
     * Functional impairment questions for late luteal phase require more than or equal to 4 score on at least one item for at least 2 or more days.
   * For women who were on anti-depressants or oral contraceptive for at least 2 months:

     * Late luteal phase daily average of 2.5 or more for at least 4 of 7 of these days on any 5 distinct items with no overlap on DRSP-scale, at least one item must represent a non-physical symptom. Entries in the diary must be present for at least three of these days for the item to be used as an inclusion criterion for that month.
     * Follicular phase daily average 2 or less for each item on DRSP scale for non-physical symptoms only. The average will be calculated for days 8-12 of the cycle, day 1 being the first day of menstrual bleeding. Entries in the diary must be present for at least three of these days for the item to be used as an inclusion criterion for that month.
     * Late luteal phase (6 days before menses through day 1 of menses) daily average at least twice as high as follicular phase daily average for three distinct items.
     * Functional impairment questions for late luteal phase require 3 or more score on at least one item for 2 or more days.
3. Absence of any one of the following Axis I disorders during the last 6 months:

   * Major Depressive Disorder
   * Anxiety Disorder (Panic Disorder, OCD, PTSD)
   * Eating Disorder
   * Drug or alcohol abuse
4. Absence of any of the following Axis I disorders (current or history of), based on the Mini International Neuropsychiatric interview (MINI)

   * Bipolar Disorder
   * Psychotic Disorder
   * Somatoform Disorder
   * Dysthymic Disorder

Other criteria:

1. Age between 18- 50.
2. Regular menstrual cycles for the 2-month period preceding enrollment into the Qualification Phase (i.e. menstrual cycle length must be between 21 and 35 days)
3. Negative Pregnancy test prior to the Treatment Phase.
4. Women must use an effective form of contraception (oral contraceptive, Barrier method, intrauterine devices, tubal ligation are considered effective forms of contraception.)
5. Judged to be in good physical health on the basis of medical history, physical examination and laboratory screening.
6. Able to understand the procedures and agree to participate in the study by signing the informed consent; in the investigator's opinion, the patient clearly intends to comply with the requirements of the study.

Exclusion Criteria:

1. Women, who are pregnant, gave birth within the last 8 months, breast-feeding or intending to become pregnant within 6 months.
2. Contraindication or hypersensitivity to levetiracetam.
3. Ongoing psychotherapy, which has begun <3months prior to the study visit.
4. Participation in another clinical trial within the last 3 months prior to the screening visit.
5. Known hypersensitivity to Levetiracetam
6. Any disease or condition that can compromise the function of body systems and which could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study medication.
7. Severe systemic disease that might interfere with the conduct of the study or the interpretation of the results.
8. Uncontrolled thyroid problems.
9. Active use of substances, excluding caffeine and nicotine, will not be permitted during the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2003-11; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Daily Record of Severity of Problems (DRSP), Clinical Global Impression- Severity (CGI-S) and Clinical Global Impression-Improvement (CGI-I). | 4 months

SECONDARY OUTCOMES:
How Levetiracetam is tolerated, adverse events. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Zerrin E Kayatekin, MD, Principal Investigator — Berkshire Medical Center
Locations (1):
- Berkshire Medical Center, Clinical Trials Program, Department of Psychiatry, Pittsfield, Massachusetts, United States